CLINICAL TRIAL: NCT06493396
Title: Effect of Opioid-free Anesthesia on Sleep Quality, Cognitive Function and Recovery Quality After General Anesthesia in Elderly Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Bijia Song, principal investigator, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: opioid-free in elderly
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Opioid-Free Anesthesia; POCD; Recovery Quality; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-free group (Experimental)
  Interventions: Drug: Opioid-free Analgesics
- Opioid group (Active Comparator)
  Interventions: Drug: Opioid group

INTERVENTIONS:
Drug: Opioid-free Analgesics — opioid free group: After infusion of a loading dose of dexmedetomidine, intravenous midazolam 2mg, propofol 2mg kg-1, esketamine 0.5 mg kg-1, rocuronium 0.6-1mg kg-1, and 3min after endotracheal intubation. Intravenous continuous infusion of propofol, esketamine and dexmedetomidine hydrochloride mixture (esketamine 50mg + dexmedetomidine hydrochloride 150 ug + 0.9% saline 50ml in the same 50ml syringe) 0.1ml kg-1 h-1-0.2 ml kg-1 h-1 (equivalent to esketamine 0.1-0.2mg kg-1 h-1; Dexmedetomidine hydrochloride 0.3-0.6 μ g kg-1 h-1) maintains a BIS value between 40-60, 10-20mg / time was added as appropriate.
  Arms: Opioid-free group
Drug: Opioid group — Intravenous midazolam 2mg, propofol 2mg kg-1, sufentanyl 0.3-0.5 μ g kg-1, rocuronium 0.6-1mg kg-1,3min before endotracheal intubation. After successful endotracheal intubation, continuous intravenous infusion of propofol and remifentanil was started to maintain BIS values between 40-60, and rocuronium 10-20mg / time as appropriate. After the start of surgery, 10-20 μ g of sufentanil was added according to blood pressure and heart rate. At the end of the operation, 5mg and 50mg were injected before the end of the operation, and propofol and remifentanil were stopped at the end of the operation
  Arms: Opioid group

SUMMARY:
Postoperative cognitive dysfunction (POCD)is a common well disorder of the central nervous system after surgery, mainly manifested by impaired memory, spirit, language ability or other aspects of brain function. POCD, which often occurs in elderly patients over 65 years, The recent phase is recommended to be changed to perioperative neurocognitive impairment ( PND), The PND is used to describe the cognitive function changes that occur before and within 1 year after surgery, Based on the time of disease onset, It can be divided into neurocognitive impairment existing before surgery, postoperative delusion (POD) occurring hours to days after surgery, neurocognitive recovery delay (DNR) within 30 days after surgery, and postoperative neurocognitive impairment occurring weeks to months after surgery (POND). With the acceleration of the aging process of Chinese social population, the frequency of surgical treatment for elderly inpatients has also increased, and the elderly patients have postoperative sleep disorders, and POCD is relatively common. Surgical patients after surgical trauma, the body inflammation, sympathetic excitation and endocrine disorders, make postoperative sleep structure or pattern change, often lead to postoperative sleep disorders (PSD) , the main performance for patients with postoperative complaint difficult to enter and maintain sleep, frequent nightmares, total sleep quantity and quality reduction, etc. PSD is not only the most common manifestation of postoperative brain dysfunction, but also an important risk factor for inducing postoperative fatigue, postoperative hyperalgesia, metabolic dysfunction, and cardiovascular and cerebrovascular diseases. Moreover, it is considered to promote the development of postoperative delusion. At present, the common mode of general anesthesia is still mainly opioids, and opioids are an important part of general anesthesia and perioperative analgesia. Perioperative use of opioids is not only associated with adverse effects such as postoperative nausea and vomiting, excessive sedation, and ileus, but also leads to the occurrence of postoperative hypoxemia, hyperalgesia and postoperative chronic pain, and cognitive impairment. Therefore, the Association of Accelerated Rehabilitation Surgery indicates that the use of a multimodal analgesic regimen during the perioperative period reduces pain and reduces opioid-related adverse effects, and that opioid-free anesthesia ( OFA) is used in clinical work. At present, most clinical studies of OFA focus on adults aged 18-65 or 18 years old, and few studies focus OFA solely on the elderly population to observe its application effect. Therefore, it is necessary to conduct clinical studies to observe postoperative recovery in elderly patients with different types of anesthetics, investigate the incidence and severity of POCD, and determine the efficacy and safety of each anesthetic agent.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients to undergo elective non-cardiac surgery

  * ASA grade I or III;

    * volunteered in this trial and signed informed consent;

      * age 60 years;

        * BMI 18-30kg / m2.

Exclusion Criteria:

* Chronic pain;

  * severe liver dysfunction (total bilirubin 2 mg dl-1);

    * severe renal dysfunction (glomerular filtration rate 60ml min-1 1.73m-2);

      * preoperative heart rate <50 beats / min, sick sinus syndrome, severe heart block;

        * dementia or significant neurological disease (such as stroke, epilepsy, intracranial tumor, Parkinson disease, etc);

          * history of alcohol or drug abuse;

            * preoperative or PSQI score 7 or sleep disturbance;

              * Cannot cooperate with the scale survey

                * Allergic to the trial drug

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
15-item recovery quality scale score 24 hours before surgery | 24 hours before surgery
  The QoR-15 scale is a global measure of postoperative recovery, with scores ranging from 0 (extremely poor QoR) to 150 (excellent QoR). QoR-15 has become the most widely reported indicator for the evaluation of postoperative life treatment in patients. Using wherever possible QoR-15 item scores on postoperative day 3, QoR-15 with very good validity, and good reliability, responsiveness and clinical acceptability, these data suggest that QoR-15 is an excellent patient-centered measure of postoperative QoR. Patient Acceptable symptom status describes the lowest absolute score considered by the patient to represent a healthy or good status health scale. A QoR-15 score of 118 or more indicates a good postoperative recovery
15-item recovery quality scale score 24 hours after surgery | 24 hours after surgery
  The QoR-15 scale is a global measure of postoperative recovery, with scores ranging from 0 (extremely poor QoR) to 150 (excellent QoR). QoR-15 has become the most widely reported indicator for the evaluation of postoperative life treatment in patients. Using wherever possible QoR-15 item scores on postoperative day 3, QoR-15 with very good validity, and good reliability, responsiveness and clinical acceptability, these data suggest that QoR-15 is an excellent patient-centered measure of postoperative QoR. Patient Acceptable symptom status describes the lowest absolute score considered by the patient to represent a healthy or good status health scale. A QoR-15 score of 118 or more indicates a good postoperative recovery
15-item recovery quality scale score 48 hours after surgery | 48 hours after surgery
  The QoR-15 scale is a global measure of postoperative recovery, with scores ranging from 0 (extremely poor QoR) to 150 (excellent QoR). QoR-15 has become the most widely reported indicator for the evaluation of postoperative life treatment in patients. Using wherever possible QoR-15 item scores on postoperative day 3, QoR-15 with very good validity, and good reliability, responsiveness and clinical acceptability, these data suggest that QoR-15 is an excellent patient-centered measure of postoperative QoR. Patient Acceptable symptom status describes the lowest absolute score considered by the patient to represent a healthy or good status health scale. A QoR-15 score of 118 or more indicates a good postoperative recovery

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index，PSQI | one night before surgery
  The PSQI scale consists of seven aspects, including time to sleep, hypnotic drugs, sleep time, daytime dysfunction, sleep quality, sleep efficiency, and sleep disorders, with a total score of 0 to 21, which is generally considered in China Score 7 means the presence of sleep disturbance, the higher the score indicates more severe sleep disturbance]; due to PSQI The simplicity of the scale has good reliability and validity, and the results of polysomnography and EEG exist larger Guan Xing, which has become the most widely used scale in sleep research at home and abroad
Pittsburgh Sleep Quality Index，PSQI | first night after surgery
  The PSQI scale consists of seven aspects, including time to sleep, hypnotic drugs, sleep time, daytime dysfunction, sleep quality, sleep efficiency, and sleep disorders, with a total score of 0 to 21, which is generally considered in China Score 7 means the presence of sleep disturbance, the higher the score indicates more severe sleep disturbance]; due to PSQI The simplicity of the scale has good reliability and validity, and the results of polysomnography and EEG exist larger Guan Xing, which has become the most widely used scale in sleep research at home and abroad
Pittsburgh Sleep Quality Index，PSQI | the second night after surgery
  The PSQI scale consists of seven aspects, including time to sleep, hypnotic drugs, sleep time, daytime dysfunction, sleep quality, sleep efficiency, and sleep disorders, with a total score of 0 to 21, which is generally considered in China Score 7 means the presence of sleep disturbance, the higher the score indicates more severe sleep disturbance]; due to PSQI The simplicity of the scale has good reliability and validity, and the results of polysomnography and EEG exist larger Guan Xing, which has become the most widely used scale in sleep research at home and abroad
Pittsburgh Sleep Quality Index，PSQI | one week after surgery
  The PSQI scale consists of seven aspects, including time to sleep, hypnotic drugs, sleep time, daytime dysfunction, sleep quality, sleep efficiency, and sleep disorders, with a total score of 0 to 21, which is generally considered in China Score 7 means the presence of sleep disturbance, the higher the score indicates more severe sleep disturbance]; due to PSQI The simplicity of the scale has good reliability and validity, and the results of polysomnography and EEG exist larger Guan Xing, which has become the most widely used scale in sleep research at home and abroad
Rhodes Index of Nausea and Vomiting | one day before surgery
  Rhodes Index of Nausea, Vomiting, and Retching, an 8-item questionnaire, to measure the incidence and severity of nausea, vomiting, and retching At each timepoint, a total Rhodes score was calculated from the sum of the 8 RINVR questions. Total Rhodes scores were compared at 6 different timepoints as well as overall across all 6 time points. record Nausea and vomiting, the Rhodes index score
Rhodes Index of Nausea and Vomiting | 6,24,48 hours after surgery
  Rhodes Index of Nausea, Vomiting, and Retching, an 8-item questionnaire, to measure the incidence and severity of nausea, vomiting, and retching At each timepoint, a total Rhodes score was calculated from the sum of the 8 RINVR questions. Total Rhodes scores were compared at 6 different timepoints as well as overall across all 6 time points. record Nausea and vomiting, the Rhodes index score
Ramsay score | 6, 24, 48 hours after surgery
  Total score: 1 to 6,1 indicates insufficient sedation and restlessness; 2 indicates quiet and cooperation; 3 indicates drowsiness and response to commands; 4 indicates shallow sleep and quick response to strong acoustic stimulation; 5 means slow to sleep and response to strong acoustic stimulation; 6 indicates too deep calm and difficult to wake up Score 7 means the presence of sleep disturbance, the higher the score indicates more severe sleep disturbance]; due to PSQI The simplicity of the scale has good reliability and validity, and the results of polysomnography and EEG are large
visual analgesia score | 6, 24, 48 hours after surgery
  The total score is 0 to 10,0 indicates no pain, and 10 indicates the most severe play ache
The Mini-Cog cognitive score | first night before surgery
  0 points: 3 words can not remember one, as dementia. 1~2 points: can remember 1~2 of 3 words, correct drawing clock test (CDT), normal cognitive function; incorrect CDT, and cognitive function deficit. 3 points: can remember 3 words, not fixed as dementia
The Mini-Cog cognitive score | first day,second day and one week after surgery
  0 points: 3 words can not remember one, as dementia. 1~2 points: can remember 1~2 of 3 words, correct drawing clock test (CDT), normal cognitive function; incorrect CDT, and cognitive function deficit. 3 points: can remember 3 words, not fixed as dementia
Number of salvage analgesia used within 48 h after surgery | 48 h after surgery
  record number of salvage analgesia used within 48 h after surgery